CLINICAL TRIAL: NCT00371735
Title: A Multi-centre, Randomised, Double-blind Study to Compare the Efficacy and Safety of Chlorproguanil-dapsone-artesunate Versus Chlorproguanil-dapsone in the Treatment of Acute Uncomplicated Plasmodium Falciparum Malaria in Children, Adolescents and Adults in Africa.
Brief Title: Chlorproguanil-Dapsone-Artesunate (CDA) Versus Chlorproguanil-Dapsone (LAPDAP) For Uncomplicated Malaria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDA 714703/006
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Malaria, Falciparum
Keywords: Malaria CDA LAPDAP Africa
MeSH Terms: conditions — Malaria, Falciparum | interventions — chloroguanil, dapsone drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: chlorproguanil-dapsone-artesunate; Drug: chlorproguanil-dapsone

INTERVENTIONS:
Drug: chlorproguanil-dapsone-artesunate
Drug: chlorproguanil-dapsone
  Other Names: chlorproguanil-dapsone-artesunate

SUMMARY:
CDA is a combination of chlorproguanil, dapsone and artesunate, being developed in a public-private partnership with the Medicines for Malaria Venture (MMV), World Health Organisation (WHO-TDR) and academic partners from the London School of Hygiene and Tropical Medicine, University of Liverpool and the Liverpool School of Tropical Medicine as a treatment for acute uncomplicated P. falciparum malaria.

The combination of chlorproguanil HCl (CPG) and dapsone (DDS) as chlorproguanil-dapsone has already been shown to be efficacious against P.falciparum in adults and children in Sub-Sahara Africa. The addition of artesunate to LAPDAP has been demonstrated to increase the parasite kill rate as demonstrated in the phase II study, and reduce the chance of any parasites escaping treatment over the 3-day course. The addition of artesunate is also anticipated to have the population benefit of protection against the development of resistant strains of P.falciparum, although it will not be possible to demonstrate this in a clinical trial. One further population benefit of the artemisinin drugs are their ability to suppress the sexual forms of the parasite (gametocytes), which should reduce infectivity after antimalarial treatment and potentially lower transmission rates with widespread use, including the spread of any parasites resistant to the partner drug.

The aims of this phase III study are to compare the efficacy of a fixed ratio combination tablet of CDA to chlorproguanil-dapsone, and collect supporting safety data. This will be a multi-centre, double-blind, double-dummy, randomised trial, in children, adolescents and adults, with chlorproguanil-dapsone as a comparator.

ELIGIBILITY:
Inclusion criteria:

* Acute, uncomplicated P.falciparum malaria, microscopically confirmed infection.
* Temperature at screening of 37.5oC or over or confirmed history of fever within previous 24-hours.
* Weight 7.5kg or over , no upper weight limit.
* Screening haemoglobin (Hb) of 7g/dl, or more or haematocrit of 25% or over(if Hb not available at screening).
* Willingness to comply with the study visits and procedures, as outlined in the informed consent form.
* Written or oral witnessed consent obtained from subject, parent or guardian.
* Assent is given by a child aged 12 to <18years, in addition to the consent of their parent or guardian.

Exclusion criteria:

* Features of severe/complicated falciparum malaria.
* Hypersensitivity to active substances (chlorproguanil, dapsone, artesunate), or excipients of the investigational products.
* Known allergy to biguanides, sulphones, sulphonamides or artemisinin derived products.
* Known history of G6PD deficiency.
* Infants with a history of hyperbilirubinaemia during the neonatal period.
* Evidence of any concomitant infection at the time of presentation (including P. vivax, P. ovale and P. malariae).
* Use of concomitant medications that may induce haemolysis or haemolytic anaemia from the WHO (World Health Organization) list of essential drugs.
* Any other underlying disease that may compromise the diagnosis and the evaluation of the response to the study medication (including clinical symptoms of immunosuppression, tuberculosis, bacterial infection; cardiac or pulmonary disease).
* Malnutrition, defined as a child whose weight-for-height is below -3 standard deviations or less than 70% of the median of the NCHS/WHO normalised reference values
* Treatment within the past three months with mefloquine or mefloquine-sulphadoxine-pyrimethamine; twenty-eight days with sulphadoxine/pyrimethamine, sulfalene/pyrimethamine, lumefantrine or artemether/lumefantrine, amodiaquine, atovaquone or atovaquone/proguanil, halofantrine; 14-days with chlorproguanil/dapsone, or 7-days with quinine (full course), proguanil, artemisinin, tetracycline doxycycline or clindamycin.
* Positive sulphadoxine/pyrimethamine urine screen for 'unknown' antimalarial drug use in prior 28-days.
* Use of an investigational drug within 30 days or 5 half-lives whichever is the longer.
* Previous participation in this study.
* Female subjects of child-bearing potential who have had a positive pregnancy test at enrolment, or do not give their consent to take a pregnancy test.
* Female subjects who will be breast-feeding an infant for the duration of the study.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2006-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Parasitological cure rate, PCR-corrected, at day 28, in the per-protocol population. Parasitological cure rate is defined as the clearance of the initial malaria infection by day 7 and remaining free of this infection to the day of assessment.

SECONDARY OUTCOMES:
The proportion of subjects with parasites remaining at 24 hours post-first dose by treatment group. Parasitological cure rate, PCR-corrected, at day 14, by treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- GSK Investigational Site, Ouagadougou, Burkina Faso
- GSK Investigational Site, Kumasi, Ghana
- GSK Investigational Site, Bamako, Mali
- Nigeria (4):
  - GSK Investigational Site, Ile-Ife
  - GSK Investigational Site, Jos
  - GSK Investigational Site, Lagos
  - GSK Investigational Site, Maiduguri

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Pamba A, Richardson ND, Carter N, Duparc S, Premji Z, Tiono AB, Luzzatto L. Clinical spectrum and severity of hemolytic anemia in glucose 6-phosphate dehydrogenase-deficient children receiving dapsone. Blood. 2012 Nov 15;120(20):4123-33. doi: 10.1182/blood-2012-03-416032. Epub 2012 Sep 19. PMID 22993389
- [Derived] Carter N, Pamba A, Duparc S, Waitumbi JN. Frequency of glucose-6-phosphate dehydrogenase deficiency in malaria patients from six African countries enrolled in two randomized anti-malarial clinical trials. Malar J. 2011 Aug 17;10:241. doi: 10.1186/1475-2875-10-241. PMID 21849081
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: CDA 714703/006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: CDA 714703/006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: CDA 714703/006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: CDA 714703/006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: CDA 714703/006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: CDA 714703/006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: CDA 714703/006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register